CLINICAL TRIAL: NCT04590313
Title: Treatment of Hallux Rigidus (HARD): A Prospective, Randomised, Controlled Trial of Arthrodesis Versus Watchful Waiting in the Treatment of Hallux Rigidus
Brief Title: Efficacy of First MTPJ Arthrodesis as a Treatment in Hallux Rigidus
Acronym: HARD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Mikko Miettinen, Consultant orthopaedic surgeon, M.D., Hospital District of Helsinki and Uusimaa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39§/30.9.2020
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Hallux Rigidus
Keywords: surgery; foot; hallux; hallux rigidus; arthrodesis
MeSH Terms: conditions — Hallux Rigidus; Ankylosis | interventions — Arthrodesis

STUDY DESIGN:
Intervention Model Description: A randomised, controlled trial will be performed by allocating 40 years or older patients with symptomatic hallux rigidus to arthrodesis or watchful waiting group in a ratio of 1:1.
Who Masked: Outcomes Assessor
Masking Description: To avoid biased interpretation of the trial data, blinded data interpretation will be used in the reporting of the results of this trial (70). Before accessing the primary outcome data, the writing committee will record a 'Background assumptions' document containing our definition of MID of the outcome measures, and a brief summary of the key statistical analysis used in the evaluation of the outcome data. The document will be signed by the members of the writing committee and published as an appendix to the primary publication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthrodesis (Active Comparator): MTPJ I Arthrodesis
  Interventions: Procedure: Arthrodesis
- Watchful waiting (No Intervention): No intervention, patient information leaflet

INTERVENTIONS:
Procedure: Arthrodesis — MTPJ I arthrodesis
  Arms: Arthrodesis

SUMMARY:
A randomised, controlled trial will be performed by allocating 40 years or older patients with symptomatic hallux rigidus to arthrodesis or watchful waiting group in a ratio of 1:1. Our primary outcome will be pain during walking, assessed by the 0-10 Numeric Rating Scale (NRS) at one year after randomisation. Our secondary outcomes will be pain in rest (NRS), physical function (MOXFQ), patient satisfaction in terms of Patient-accepted Symptom State (PASS), health-related quality of life (EQ-5D-5L), activity level (The Foot and Ankle Ability Measure Sports subscale), use of analgesics or orthoses and rate of complications. Our null hypothesis is that there will be no difference between arthrodesis and watchful waiting in treatment of hallux rigidus. Our primary analysis will be done using intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or over
* Diagnosis of hallux rigidus: Persistent pain on movement of the first MTPJ AND Osteoarthritic first MTPJ in plain X-rays
* Duration of symptoms ≥1 year
* Pain-NRS during walking of 4 or more on a scale 0-10 (higher is worse)
* No substantial pain in other joints of the foot in clinical examination
* Willingness to accept both treatment options
* Ability to understand trial information and answer outcome assessments in Finnish
* Signed informed consent

Exclusion Criteria:

* ASA* physical status classification level III or higher
* Patients with weak co-operation (dementia, schizophrenia, etc.)
* Patients with neuropathy, i.e. unable to feel 10g monofilament pressure in less than 8 out of 10 standard testing sites
* Active bacterial infection or ulcer of the lower limb
* Diabetes mellitus with insulin treatment
* Diabetes mellitus and GHb-A1C >64 mmol/mol (regardless of treatment)
* History of rheumatoid arthritis, gout or other inflammatory arthritis of the foot
* Hallux valgus angle >15° in weight-bearing X-ray
* Hallux varus in weight-bearing X-ray
* Large bone cysts in X-ray probably requiring bone grafting in surgery
* Pain in passive manipulation of ipsilateral first toe IP joint
* Patients with severe circulatory disorder of the lower limb: absence of palpable pulses in the foot (both dorsalis pedis artery and tibialis posterior artery)
* History of surgery of the foot in question
* Neuropathic pain of the foot in question (i.e., use of neuropathic analgesics)
* Activity limiting symptoms from an earlier fracture or ligament injury of the foot
* Patient is not willing to accept the operation within the planned time limits (3 to 12 weeks post-randomisation)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-06-04 (Estimated); Study Completion 2029-06-04 (Estimated)

PRIMARY OUTCOMES:
Pain during walking in Numerical Rating Scale (NRS) | 1 year after randomisation
  scale 0-10; 0=no pain, 10=worst pain

SECONDARY OUTCOMES:
Pain during rest in Numerical Rating Scale (NRS) | 6 months, 1year, 2 years, 5 years
  scale 0-10; 0=no pain, 10=worst pain
Pain during walking in Numerical Rating Scale (NRS) | 6 months, 2 years, 5 years
  scale 0-10; 0=no pain, 10=worst pain
Patient Related Outcome | 6 months, 1year, 2 years, 5 years
  MOXFQ-score, Scale 0-100
Patient reported quality of life | 6 months, 1year, 2 years, 5 years
  EQ-5D-5L, Scale 0-100
Complications | 6 months, 1year, 2 years, 5 years
  Number of minor and major adversary effects
Patient Acceptable Symptom State | 6 months, 1year, 2 years, 5 years
  Percentage of patients with acceptable symptom state (PASS)
Patients physical activity | 6 months, 1year, 2 years, 5 years
  FAAM Sports Subscale, Scale 0-100
Use of analgesics and orthoses | 6 months, 1year, 2 years, 5 years
  The use of analgesics: 1) no use of analgesics or less frequent than weekly, 2) weekly use of analgesics, 3) daily use of NSAIDS or paracetamol, 4) daily use of opioids.
  The use of orthoses: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Repo, M.D., Ph.D., Study Director — Hospital District of Helsinki and Uusimaa
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miettinen M, Ramo L, Lahdeoja T, Sirola T, Sandelin H, Ponkilainen V, Repo JP. Treatment of hallux rigidus (HARD trial): study protocol of a prospective, randomised, controlled trial of arthrodesis versus watchful waiting in the treatment of a painful osteoarthritic first metatarsophalangeal joint. BMJ Open. 2021 Aug 27;11(8):e049298. doi: 10.1136/bmjopen-2021-049298. PMID 34452964